CLINICAL TRIAL: NCT04228705
Title: Study on Comprehensive Strategy of Perioperative Pain Prevention and Treatment in Elderly Patients -- Establishment and Validation of Early-warning Model of Perioperative Pain for the Elders
Brief Title: Establishment and Validation of Early-warning Model of Perioperative Pain for the Elders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Zhejiang University (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Director of department of anesthesiology and pain management, Peking University People's Hospital
Other Study IDs: 2019PHB258-01
Record Dates: First submitted 2020-01-12; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Pain; Pain Assessment; Elderly; Model
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The elders: Patients aged over 59 years old
- The young adults: Patients aged from 18 to 59 years old

SUMMARY:
This study will collect perioperative pain-related data of elderly patients in multi-centers. Analyzing these collected data to find the high-risk factors of postoperative pain in elderly patients and to establish an early-warning model of perioperative pain in elderly patients, so as to improve the ability of assessing the risks of postoperative pain in elderly patients and providing an early warning.

DETAILED DESCRIPTION:
This study will collect perioperative pain-related data of elderly patients in multi-centers, including: preoperative general data, intraoperative anesthesia and surgical data, clinical laboratory data, postoperative pain and intervention, postoperative complications and quality of life. Analyzing these collected data to find the high-risk factors of postoperative pain in elderly patients and to establish an early-warning model of perioperative pain in elderly patients, so as to improve the ability of assessing the risks of postoperative pain in elderly patients and providing an early warning.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing general or regional anesthesia
* Hospitalized for at least 24 hours after surgery
* Able to give informed consent
* Able to read and write

Exclusion Criteria:

* Existing diagnoses of psychiatric or neurologic pathology
* A history of substance abuse
* Admitted to ICU after surgery
* Patients with advanced tumors who have received preoperative chemotherapy or who are expected to receive postoperative chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older undergoing general or regional anesthesia of any procedures, mainly include: breast surgery, thoracic surgery, abdominal surgery, total knee or hip replacement surgery and spine surgery.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-12-12 (Estimated); Study Completion 2020-12-12 (Estimated)

PRIMARY OUTCOMES:
Pain trajectories after surgery | within 6 months
  The pain trajectory is the vector of mean pain severity domain score (from 0 to 10) measured with pain severity domain of the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R)
Pain trajectories after surgery | within 6 months
  The pain trajectory is the vector of mean pain severity domain score (from 0 to 10) measured with Brief Pain Inventory -Short Form (BPI-SF) within 6 months

SECONDARY OUTCOMES:
Outcome of 6-mins-walking test | 1, 3, 7, 14, 21, 30, 60, 90, 120, 150 and180 days postoperation
  Walking distance of 6 minutes
Postoperative duration of stay in hospital | 30 days postoperation
  The duration when patients stay in hospital after surgery.
Number of readmission within 30 days after surgery | Up to 30 days postoperation
  Readmission indicates unplanned readmission after hospital discharge.
Complications within 30 days after surgery | Up to 30 days postoperation
  Complications within 30 days after surgery will be classified using Clavien-Dindo Classification of Surgical Complications, ranging from Grade I(Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions) to Grade V(death of a patient).
The trajectories of health related quality of life(HRQoL) | 1, 3, 7, 14, 21, 30, 60, 90, 120, 150 and180 days postoperation
  The trajectory of HRQoL is the vector of Utility values measured with EuroQol five-dimensional questionnaire(EQ-5D)taken over 6 months(days 1, 3, 7,14, 21, 30, 60, 90, 120, 150,180; Day 0 is the day of surgery). The EQ-5D measures health on five domains (mobility, self-care, usual activities, pain discomfort, and anxiety-depression), and the scores will be combined using Chinese general population weights to generate a single utility or index score. Utility values for the EQ-5D range from 1.00 to -0.391, where a score of 0 and 1 are regarded as equivalent to death and 'perfect health', respectively, and a score < 0 is considered as health state that is 'worse than death'.
Ambulation time | Up to 30 days postoperation
  The first time when patients can get off of bed and walk after surgery
Oral feeding time | Up to 30 days postoperation
  The first time when patients begin oral feeding after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Feng Yi, MD, PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China